CLINICAL TRIAL: NCT05927194
Title: Evaluation of Using the Connect: A Game-Based Intervention for Adolescent Pregnancy Prevention
Brief Title: Using the Connect: Game Based Intervention
Acronym: UTC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Texas A&M University (Other)
Responsible Party: Principal Investigator, Brittany Rosen, Research Associate Professor, Children's Hospital Medical Center, Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-0471
Record Dates: First submitted 2023-06-06; First posted 2023-07-03 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2024-08

CONDITIONS: Adolescent Behavior; Contraception; Health Behavior
Keywords: Adolescent Pregnancy Prevention; Sexual Health Education
MeSH Terms: conditions — Adolescent Behavior; Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Using the Connect (Experimental): Using The Connect (UTC) is a game-based learning program designed for middle school-aged youth (ages 9-15 or grades 6-8) consisting of four games played in a facilitated environment, and one take-away activity. The goals of the program include:To be a vehicle that encourages community sharing of healthy teen behavior. To facilitate safe connections between youth and adults in their community. To empower youth to lead healthy sexual lives. The four games each focus on specific health content or skills including growth and development, accessing information, positive communication, and decision-making. Each of the four games is intended to be played for a total of 90 minutes, split up into sessions of 30 minutes per game. When combining all gameplay sessions, along with the instructions for the take-away activity and program wrap-up activity, organizations will dedicate approximately 8 hours to the program.
  Interventions: Behavioral: Using the Connect
- Business as Usual (No Intervention): Participants will not receive the Using the Connect curriculum.

INTERVENTIONS:
Behavioral: Using the Connect — Using the Connect (UTC) is an innovative, game-based intervention for youth to develop skills in adulthood preparation topics such as communication, decision making and accessing information.
  Arms: Using the Connect

SUMMARY:
The study aims to implement Using the Connect (UTC), an innovative, game-based intervention designed to increase protective factors and decrease adolescent pregnancies. This intervention will be implemented in Texas middle schools and community-based organizations. The long-term goal is to promote optimal health in youth and prevent adolescent pregnancy in populations disproportionately impacted by adolescent pregnancy and sexually transmitted infection (STI) rates. The short-term objective is to conduct a robust, multi-site clustered randomized controlled trial to evaluate implementation outcomes and the impact of UTC, a novel theory-based game developed using powerful and effective human-centered design (HCD) strategies, on intention to delay sexual activity.

DETAILED DESCRIPTION:
Background: While the teen birth rate for the US is at a historic low of 16.7 per 1000 females, the state of Texas ranks 5th in teen pregnancies and 7th in teen births. The teen birth rate for the state of Texas is 22.4 per 1000 females.

Using the Connect (UTC) is an innovative, game-based intervention for youth designed by youth and community stakeholders to increase protective factors and decrease adolescent pregnancies. UTC enhances the learning environment and can be implemented in various settings including classrooms, after-school programs, community-based organizations, and with other youth age groups. Interventions developed by youth that are adaptable to meet community context and needs are lacking. UTC is a youth-developed intervention formatively tested with positive results and acceptability in areas of North Carolina and Texas. Specifically, the formative evaluations results showed that youth found the design of UTC highly acceptable, felt the games and content were engaging and relatable, and learned knowledge and skills around adolescent development, accessing information, communication, and making healthy decisions through playing the games. Youth participants reported that they would recommend the program to friends, would participate in the program again, and use the information they learned from the program in the future. The game-based program offers knowledge and skill development in adulthood preparation subjects including communication, decision making, and accessing information. In addition, the game is engaging and provides opportunities for peer interaction. This innovative intervention changes the environment that facilitators and youth are often presented in adolescent health programs and offers an interesting and unique opportunity for skill development and community building.

Purpose: The purpose of this study is to conduct a multi-site clustered randomized controlled trial to evaluate the impact of UTC, a novel theory-based game developed using powerful and effective human-centered design (HCD) strategies, on intention to delay sexual intercourse.

The primary research question:

1. How does UTC impact youth's intention to delay sexual intercourse, compared to youth who have not received UTC, at post-test and 3-month follow-up?

Methods: A multi-site clustered randomized controlled trial will be conducted to determine the effectiveness of UTC on primary outcomes. A combination of school sites and community-based organization sites will be recruited and randomized to serve as either a treatment or control group. Up to 1,800 participants will complete validated surveys at baseline (prior to participating in the treatment or control group) and immediate post (after participating in the treatment or control group), followed by 3-month, and 9-month follow-up surveys. The surveys will be approximately 30-minutes long.

Implications:

Primary Research Question:

1. How does UTC impact youth's intention to delay sexual intercourse, compared to youth who have not received UTC, at post-test and 3-month follow-up?

ELIGIBILITY:
Inclusion Criteria:

* Middle school-aged youth at one of the participating community-based organization or school sites in Texas
* Ability to complete Using the Connect in English
* Ability to read and complete surveys in English without assistance

Exclusion Criteria:

* Unable to read and speak in English

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1400 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in youth's intention to delay sexual intercourse before Using the Connect to 3 months post Using the Connect via self-reported questionnaire. | 3-months
  How does UTC impact youth's intention to delay sexual intercourse, compared to youth who have not received UTC at 3-month follow-up?

CONTACTS AND LOCATIONS:
Overall Officials: Brittany Rosen, PhD, MEd, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No